CLINICAL TRIAL: NCT01355328
Title: Evaluating Light-tissue Reaction and Transdermal Drug Delivery by Multiphoton Microscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Other Study IDs: 97105
Record Dates: First submitted 2010-05-24; First posted 2011-05-18 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2009-02

CONDITIONS: Healthy
Keywords: light
MeSH Terms: interventions — Lasers

ARMS (2):
- laser (Experimental)
  Interventions: Procedure: laser and radiofrequency
- control (No Intervention)

INTERVENTIONS:
Procedure: laser and radiofrequency — different laser and radiofrequency with different fluences
  Other Names: drug penetration
  Arms: laser

SUMMARY:
In this study, the investigators will evaluate the potential of multiphoton microscopy as a non-invasive imaging modality for monitoring of the radiofrequency-tissue and light-tissue reaction. The investigators will also investigate drug delivery using multiphoton microscopy.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults

Exclusion Criteria:

* younger than 18 years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2009-02; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Taipei, Taipei, Taiwan